CLINICAL TRIAL: NCT05956366
Title: Effectiveness of Family-based Intervention in a Child and Adolescent Mental Health Service for Children and Adolescents With Eating Disorders
Brief Title: Effectiveness of Family-based Intervention for Youn Persons With Eating Disorders
Acronym: VIBUS-wp1
Status: Recruiting | Type: Observational
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-17022391
Record Dates: First submitted 2023-02-02; First posted 2023-07-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Eating Disorders
Keywords: eating disorders, adolescents
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorexia nervosa: Children and adolescents presenting for treatment for anorexia nervosa typica or atypica (ICD-10: F50.0 or F50.1)
  Interventions: Behavioral: Family-based treatment
- Bulimia nervosa: Children and adolescents presenting for treatment for bulimia nervosa typica or atypica (ICD-10: F50.2 or F50.3)
  Interventions: Behavioral: Family-based treatment
- Other eating disorders: Children and adolescents presenting for treatment for other eating disorders (ICD-10: F50.8)
  Interventions: Behavioral: Family-based treatment

INTERVENTIONS:
Behavioral: Family-based treatment — Open-end family therapy ad modum The Maudsley model
  Other Names: FBT

SUMMARY:
This research project aims to characterize a naturalistic cohort of children and adolescents with eating disorders in terms of biological, psychological and psychopathological features. Further, the project will examine the effectiveness of treatment, the determinants of treatment outcome and the course of treatment response for children and adolescents with eating disorders (ED), treated in a generic specialist child and adolescent mental health service. The first choice of treatment is outpatient family-based treatment (FBT), which has documented effect for anorexia nervosa and bulimia nervosa. However, a subgroup of young persons with eating disorders does not respond sufficiently to this treatment, and evidence concerning effective treatment for children and adolescents with atypical eating disorders is still lacking. Further, treatment effectiveness for children and adolescents in a Danish naturalistic setting has never been examined.

DETAILED DESCRIPTION:
The overall aim is to assess associations between patient characteristics and treatment response across the spectrum of eating disorders to identify, which patients benefit from family based treatment, and which patients possibly would need other kinds of treatment or more intensive care.

Research questions:

1. Which patient and family characteristics predict faster recovery from ED in childhood and adolescence?
2. Which patient and family characteristics predict intensification of treatment in the forms of day hospital or full hospitalization?
3. At which time point can recovery be predicted based on information from initial assessment and/or assessment during the course of treatment?
4. Which patient and family characteristics (e.g. patterns of comorbid symptoms) are common in those not responding well to treatment within each diagnostic category?
5. How many young patients migrate between ED diagnoses, and what characterizes these patients?
6. Studies on treatment effectiveness for EDNOS in children and adolescents are still lacking. Hence, an important research question of this study is whether family based treatment for EDNOS is effective and is perceived as helpful by patients and families?

   In addition, the project will seek to answer the following:
7. Is treatment effectiveness in The Capital Region of Denmark (BUC) comparable to published results from other countries in the same age group?

ELIGIBILITY:
Inclusion Criteria:

* begin treatment for eating disorder

Exclusion Criteria:

* lack of informed consent

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients assessed and treated for any eating disorder (ICD-10: F50.0-F50.8) in the unit for treatment of eating disorders will be invited to participate.
  Due to the naturalistic design of this study we will examine a representative, consecutive sample, without any exclusion criteria except the absence of informed consent by patient and parents or legal care takers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of participants with weight normalisation | through treatment completion an average of 1 year
  at or above 95% of ideal BMI adjusted for age and gender, based on the individual´s prior growth trajectory. BMI is calculated as weight in kg/(height in meters*height in meters), and percentage if ideal BMI adjusted for age and gender is based on published, standardized growth curves from Danish children and adolescents
proportion of participants with weight normalisation | 2.5 years after treatment completion
  at or above 95% of ideal BMI adjusted for age and gender, based on the individual´s prior growth trajectory. BMI is calculated as weight in kg/(height in meters*height in meters), and percentage if ideal BMI adjusted for age and gender is based on published, standardized growth curves from Danish children and adolescents
proportion of participants with weight normalisation | 5 years after treatment completion
  at or above 95% of ideal BMI adjusted for age and gender, based on the individual´s prior growth trajectory. BMI is calculated as weight in kg/(height in meters*height in meters), and percentage if ideal BMI adjusted for age and gender is based on published, standardized growth curves from Danish children and adolescents
proportion of participants with weight normalisation | 7.5 years after treatment completion
  at or above 95% of ideal BMI adjusted for age and gender, based on the individual´s prior growth trajectory. BMI is calculated as weight in kg/(height in meters*height in meters), and percentage if ideal BMI adjusted for age and gender is based on published, standardized growth curves from Danish children and adolescents
proportion of participants with weight normalisation | 10 years after treatment completion
  at or above 95% of ideal BMI adjusted for age and gender, based on the individual´s prior growth trajectory. BMI is calculated as weight in kg/(height in meters*height in meters), and percentage if ideal BMI adjusted for age and gender is based on published, standardized growth curves from Danish children and adolescents
proportion of participants with absence of eating disordered behaviors | through treatment completion an average of 1 year
  absence for 4 weeks (according to diagnostic questions if Eating Disorder Examination (EDE).
proportion of participants with absence of eating disordered behaviors | 2.5 years after treatment completion
  absence for 4 weeks (according to diagnostic questions if Eating Disorder Examination (EDE).
proportion of participants with absence of eating disordered behaviors | 5 years after treatment completion
  absence for 4 weeks (according to diagnostic questions if Eating Disorder Examination (EDE).
proportion of participants with absence of eating disordered behaviors | 7.5 years after treatment completion
  absence for 4 weeks (according to diagnostic questions if Eating Disorder Examination (EDE).
proportion of participants with absence of eating disordered behaviors | 10 years after treatment completion
  absence for 4 weeks (according to diagnostic questions if Eating Disorder Examination (EDE).

CONTACTS AND LOCATIONS:
Overall Officials: Mette Bentz, PhD, Principal Investigator — Child and Adolescent Mental Health Care Centre, Capital Region of Denmark; Anne Katrine Pagsberg, professor, Study Director — Child and Adolescent Mental Health Care Centre, Capital Region of Denmark
Locations (1):
- Child and Adolescent Mental Health Care Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bentz M, Pedersen SH, Moslet U, Petersen N, Pagsberg AK. Predictors of response to family-based treatment for anorexia nervosa in youth: insights from the VIBUS project. Eur Child Adolesc Psychiatry. 2025 Nov;34(11):3665-3684. doi: 10.1007/s00787-025-02766-x. Epub 2025 Jun 11. PMID 40498327